CLINICAL TRIAL: NCT04053725
Title: A Prospective Study of Blood Circulating Tumor DNA for the Prediction of Efficacy in Immunotherapy for Advanced Gastric Cancer.
Brief Title: Prediction of the Efficacy of ctDNA in Immunotherapy for Advanced Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, president, Sun Yat-sen University
Other Study IDs: SYSUCC-ctDNA
Record Dates: First submitted 2019-06-16; First posted 2019-08-12 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Gastric cancer is one of the common malignant tumors in China, with relatively high incident rate and mortality among the population. Surgery is the conventional treatment option for early and intermediate-stage stage gastric cancer, but postoperative relapse is the major issue. Circulating tumor DNA (ctDNA) is tumor-derived fragmented DNA with an average size of 166 bp, mixed with cell free DNA (cfDNA) of other sources in blood circulation.ctDNA is reflecting the most up-to-date status of tumor genome. Hence, it is considered as a new biomarker for tumor, which can be qualitative, quantitative and used for disease monitoring. The present clinical trial aims to explore the possibility of clinical utility of serum ctDNA as a clinical index to predict the efficacy in immunotherapy for advanced gastric cancer.

DETAILED DESCRIPTION:
Gastric cancer is one of the most common malignant tumors in China, with the second highest incidence and the third highest mortality.Adenocarcinoma accounts for 95% of gastric malignancies and is the most common malignancy of the digestive tract. Seventy percent of the patients with early gastric cancer had no obvious symptoms, and a few had nausea, vomiting or ulcer-like upper gastrointestinal symptoms.

Surgical treatment is the first choice for the treatment of early gastric cancer, but postoperative recurrence and metastasis are prone to occur. At the same time, there are relatively few chemotherapy drugs for gastric cancer, only a few chemotherapy drugs of Paclitaxel and platinum drugs are selected, and the chemotherapy regimen is relatively single. Meanwhile, the prognosis of gastric cancer in different parts is significantly different, and its molecular heterogeneity is strong. Studies have shown that about 13% of gastric cancer has HER2 gene variation, and there is no other specific driver gene mutation except HER2. Currently, only two targeted drugs, trastuzumab and apatinib, are approved for the treatment of gastric cancer in China.

CtDNA is the body's endogenous tumor DNA free of cells in circulating blood. It is generally believed that ctDNA in the blood of tumor patients is mainly derived from tumor cell necrosis and proliferation after apoptosis, as well as the release of proliferative and active tumor cells. At present, most studies have proved that the DNA of tumor cells has consistent genetic changes with ctDNA, and the same genetic changes may be detected in the plasma free DNA of patients with driver gene mutations in the primary or metastatic lesions. Therefore, ctDNA is a characteristic tumor biomarker and can be qualitatively, quantitatively and dynamically tracked.

Immunoassay point inhibitors, including pd-1 inhibitors, pd-l1 inhibitors and ctla-4 inhibitors, have achieved significant efficacy in a variety of tumors and are expected to change the treatment status of tumors. In the case of gastric cancer, recently the Lancet Oncology published the final results and review of the KEYNOTE 012 study that investigated the efficacy of Pembrolizumab in patients with advanced pd-l1 positive gastric cancer. Results showed that 53% of patients had tumor regression, 22% had partial imaging remission, and the median duration of remission was 40 weeks. Pembrolizumab is also superior to standard second-line chemotherapy. However, currently there is no recognized indicator that can predict the efficacy of immunotherapy for gastric cancer, and relevant research is urgently needed.

The purpose of this study was to investigate the correlation between the dynamic changes of ctDNA during surgery and the effect of immunotherapy on gastric cancer patients and its effect as a hematological index for the prognosis of advanced gastric cancer. Meanwhile, molecular markers related to the prognosis of advanced gastric cancer were screened out by comparing the differences in the molecular characteristics of gastric cancer tissues among patients with different prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age at first visit.
2. Patients must have histologically confirmed gastric cancer .
3. Patients were surgically assessed to be inoperable.
4. Patients received second-line or third-line chemotherapy and were treated with immunoassay point inhibitors.
5. Patients' early pathological information was complete, including tumor site and pathological type.
6. Patients must be able to provide sufficient fresh tissue/biopsies or minimum 5-10 FFPE sections for NGS analysis.
7. Patients must be able to follow the study visit schedule and willing to provide peripheral blood samples at the indicated time point.
8. Written informed consent must be obtained from patient or patient's legal representative and ability for patient to comply with the requirements of the study.

Exclusion Criteria:

1. Patients who cannot provide peripheral blood samples prior to the surgical treatment will be excluded.
2. Patients with severe infection will be excluded.
3. Patients with other serious disease besides gastric cancer will be excluded.
4. Pregnant women will be excluded.
5. Patients who are alcoholic or drug abusers will be excluded.
6. Patients with a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data will be excluded.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This prospective clinical study program enrolled 80 patients. Patients should be treated with second- or third-line chemotherapy and combined with immunoassay inhibitors. The pre-treatment plasma ctDNA sample mutation information of each patient was compared with the tissue sample mutation information. The pre-treatment ctDNA dynamic monitoring results were compared with the ctDNA mutation information after treatment initiation. The post-treatment ctDNA dynamic monitoring results and imaging comparison analysis.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
the proportions of patients with positive serum ctDNA that have postoperative relapse | through study completion, an average of 2 years
  the proportions of patients with positive serum ctDNA (in any follow-up) that have postoperative relapse

SECONDARY OUTCOMES:
The proportion of ctDNA content decreased in patients with good therapeutic effect | through study completion, an average of 2 years
  The proportion of patients with good therapeutic effect whose serum ctDNA content decreased (in any follow-up）

CONTACTS AND LOCATIONS:
Overall Officials: Rui-hua Xu, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer center of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided